CLINICAL TRIAL: NCT06783725
Title: Improving Sleep and Quality of Life in Individuals with Down Syndrome and Their Caregivers
Brief Title: Sleep Intervention and Quality of Life in Down Syndrome
Acronym: SleepDS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Caroline G. Richter, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300013331; 3128827.000.213128827.48160000 (Other: University of Alabama at Birmingham)
Record Dates: First submitted 2024-12-27; First posted 2025-01-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Down Syndrome; Down Syndrome (Trisomy 21)
Keywords: Down syndrome; sleep; Mindfulness-Based Therapy for Insomnia
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mindfulness-Based Therapy for Insomnia (Experimental): Individuals with Down syndrome will receive the MBTI intervention over 8 sessions lasting 1 hour over 8 weeks (one session per week). One trained graduate research assistant will deliver the intervention with supervision of a licensed Clinical Psychologist.
  Interventions: Behavioral: Mindfulness-Based Therapy for Insomnia
- Wait-list control (Placebo Comparator): The control group will do the pre and post assessments but will not be part of any intervention. The wait-list control group will receive the MBTI intervention after the post-intervention measures are completed.
  Interventions: Behavioral: Wait-list control

INTERVENTIONS:
Behavioral: Mindfulness-Based Therapy for Insomnia — Mindfulness-based therapy for insomnia (MBTI) is a structured program designed to help individuals with chronic insomnia improve their sleep patterns through mindfulness practices. It combines mindfulness meditation, cognitive behavioral strategies, and sleep education to address the cognitive and physiological factors that disrupt sleep. The therapy emphasizes present-moment awareness, acceptance of sleep difficulties, and the reduction of sleep-related anxiety to promote better sleep quality and overall well-being.
  Arms: Mindfulness-Based Therapy for Insomnia
Behavioral: Wait-list control — The wait-list control group consists of participants who do not receive the intervention during the initial study period but are placed on a waitlist to receive it after the trial concludes. This group serves as a comparison to evaluate the effectiveness of the intervention while ensuring participants eventually have access to the treatment. It helps control for natural changes over time and the psychological effects of expecting future treatment.
  Arms: Wait-list control

SUMMARY:
Aim 1 of the proposed project will be to adapt the virtual Mindfulness-Based Therapy for Insomnia (MBTI) for individuals with Down syndrome (DS). The investigators will work closely with a community advisory board consisting of individuals with DS, their caregivers, and clinicians specializing in DS and sleep medicine to ensure that the intervention protocol is relevant and appropriate for young people with DS (age 12 and older). Planned adaptations include 1) utilization of visual aids and videos to increase engagement and reinforce mindfulness concepts and practices; 2) shortened meditation practices to accommodate concentration limits of individuals with DS; 3) caregiver involvement reflecting the important role of caregivers in daily functioning of individuals with DS; 4) adapted homework to cater to the learning styles of individuals with DS; 5) daily reminders to encourage regular practice and reinforce the importance of consistency; and 6) modified session structure to ensure that participants are able to discuss their experiences and refine their mindfulness practice. During the first 6 months of the project, the investigators will meet monthly with the community advisory board and use an iterative process to develop detailed intervention protocol for a virtual MBTI suitable for young people with DS.

Aim 2 of the project will be to pilot test the efficacy of the virtual MBTI for young people with DS. In the second half of the one-year project, the investigators will conduct a pilot randomized clinical trial (RCT) of the intervention developed in Aim 1.

This project will compare the effectiveness of Mindfulness Based Therapy for Insomnia (MBTI) and Brief Behavioral Therapy for Insomnia (BBTI) for young people with Down syndrome (DS). The interventions will be compared on their impact on improving sleep problems, quality of life, and functional outcomes. This project will also test if targeting the sleep of the caregiver in addition to the individual with Down syndrome has any effect on the outcomes.

DETAILED DESCRIPTION:
This study aims to address the significant gap in effective behavioral treatments for sleep problems in individuals with Down syndrome (DS). Specifically, it focuses on testing the efficacy of a virtual Mindfulness-Based Therapy for Insomnia (MBTI) for individuals with DS aged 12-30 years, along with their caregivers. The intervention seeks to improve sleep quality and overall quality of life for both participants and their caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a confirmed diagnosis of Down syndrome (DS).
* English is the primary language spoken in the household.
* Nonverbal mental age of at least 36 months, as determined by a baseline measure of adaptive skills.
* Presence of at least one sleep disturbance occurring five or more nights per week, as reported by a caregiver. Sleep disturbances may include: Bedtime resistance; Delayed sleep onset; Problematic sleep associations; Nighttime awakenings; Early morning awakenings

Exclusion Criteria:

* Severe sensory or motor impairments that would interfere with participation in the intervention.
* Inability to complete assessments or participate in the intervention sessions due to behavioral or medical conditions.
* Participation in other concurrent behavioral or sleep interventions.
* Caregiver inability or unwillingness to provide accurate reports or assist in intervention activities as needed.

Ages: 12 Months to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Sleep Quality - Sleep duration | Before (week 0) and at week 9 (the end of the 8-week intervention period).
  Assessed using wearable devices (FitBit Versa 4), which record sleep parameters: Sleep duration (in hours).
  Sleep duration in hours will be averaged over seven consecutive days, before and after the 8-week intervention.
  Higher scores indicate better outcome.
Objective Sleep Quality - Sleep efficiency | Before (week 0) and at week 9 (the end of the 8-week intervention period).
  Assessed using wearable devices (FitBit Versa 4), which record sleep parameters: Sleep efficiency (percentage of time spent asleep while in bed).
  Higher scores indicate better outcome.
Objective Sleep Quality - Number of night awakenings | Before (week 0) and at week 9 (the end of the 8-week intervention period).
  Assessed using wearable devices (FitBit Versa 4), which record sleep parameters: Number of night awakenings (count for night awakenings)
Subjective Sleep Quality - Children's Sleep Habits Questionnaire | Before (week 0) and at week 9 (the end of the 8-week intervention period).
  Measured using standardized parent-reported questionnaires:
  - Children's Sleep Habits Questionnaire (CSHQ): Assesses sleep behaviors and patterns. The CSHQ is a retrospective, 45-item parent questionnaire.
  Scale Range: 45-135. Higher scores indicate worse sleep quality. Unit of Measure: Raw score
Subjective Sleep Quality - Insomnia Severity Index | Before (week 0) and at week 9 (the end of the 8-week intervention period).
  - Insomnia Severity Index (ISI): Measures the severity of insomnia symptoms. Scale Range: 0-28. Higher scores indicate worse insomnia severity.

SECONDARY OUTCOMES:
Quality of life - Caregiver report | Before (week 0) and at week 9 (the end of the 8-week intervention period).
  Quality of life is a secondary outcome variable, evaluated using caregiver-reported measures: 1) Pediatric Quality of Life Inventory (PedsQL): Assesses health-related quality of life across physical, emotional, social, and school functioning domains. Scale Range: 0-100. Higher scores indicate better quality of life. Changes in scores before and after the intervention will be compared to evaluate improvements in quality of life.
Quality of life | Before (week 0) and at week 9 (the end of the 8-week intervention period).
  Quality of life is a secondary outcome variable, evaluated using caregiver-reported measures:
  2) KidsLife: Measures quality of life specific to individuals with developmental disabilities, including participation and independence. Scale Range: 0-100. Higher scores indicate better quality of life.
Quality of life | Before (week 0) and at week 9 (the end of the 8-week intervention period).
  Quality of life is a secondary outcome variable, evaluated using caregiver-reported measures:
  3) KIDSCREEN-27: Evaluates physical well-being, psychological well-being, autonomy, social support, and peer relationships. Scale Range: 0-100. Higher scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline G Richter, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No